CLINICAL TRIAL: NCT02811224
Title: Ovarian Cancer Hemoscope Trial
Status: Active, not recruiting | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 15-6644
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ovarian Cancer
- Benign Neoplasm

SUMMARY:
This is a prospective, gold standard observational trial designed to enroll consecutive, consenting ovarian cancer patients for the purpose of determining sensitivity of an assay that detects circulating tumor DNA. This observational pilot trial will also be used to examine the genetic variants/mutations present in the tumor tissue DNA.

ELIGIBILITY:
Inclusion Criteria:

Case Group

* Patients with ovarian cancer undergoing surgery (all stages)
* Over 18 years old

Control Group

* Patients with a benign gynecological condition undergoing surgery
* Over 18 years old

Exclusion Criteria:

* Previous cancer diagnosis (all)
* Radiation therapy before surgical treatment
* Bone marrow transplant
* Chemotherapy before surgical treatment
* Invasive procedure resulting in damage to tissue (e.g., surgery, biopsy, thermal ablation) in the 7 days prior to baseline (pre-surgical) blood collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing surgery as part of the treatment plan for ovarian cancer or a benign gynecological neoplasm.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-05; Primary Completion 2025-06 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of an assay that detects circulating tumor DNA | 3 years

IPD SHARING:
Plan to Share IPD: Undecided